CLINICAL TRIAL: NCT03074084
Title: Acute Abdomen in Adults- a Prospective Study on Causes of Abdominal Pain Leading to Emergency Department Admission in Tampere University Hospital
Brief Title: Acute Abdomen in Adults- a Prospective Study on Emergency Department Admissions
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tampere University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: R16006
Record Dates: First submitted 2016-10-20; First posted 2017-03-08 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Abdominal Pain
Keywords: abdominal pain; adult; emergency department; electronic nose; celiac disease
MeSH Terms: conditions — Abdominal Pain; Emergencies; Celiac Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — urine sample, blood sample
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a non-randomized, prospective, population-based, single-center study designed to evaluate conditions resulting emergency admission in patients with abdominal pain. Furthermore, we are interested in how many patients are discharged with "non-specific abdominal pain" but later readmitted and diagnosed with a specific diagnosis.

DETAILED DESCRIPTION:
1000 adult patients with acute abdominal pain will be recruited at Tampere University Hospital Emergency department. The patients will fill in a questionaire about the symptoms and their duration. A urine sample will be collected for polyamine molecule analysis with an electronic nose. At later stage of the study, a serum sample for coeliac tests will be collected. Patient outcome will be obtained during the hospital stay, at one-month after discharge and at one year.

ELIGIBILITY:
Inclusion Criteria:

All adult patients with abdominal pain.

Exclusion Criteria:

Under the age of 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the adult patients with abdominal pain admitted to the emergency department are included. One thousand patients from Tampere district will be chosen for analysis.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-06; Primary Completion 2021-12 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with specific diagnose | One month
  Population based analysis of incidence of diseases

SECONDARY OUTCOMES:
Number of patients misdiagnosed in emergency department and requiring readmission | One month
Number of participants with treatment related adverse events | One month
Diagnostic accuracy of polyamine molecule analysis | One month
Number of patients with undiagnosed coeliac disease | One month

CONTACTS AND LOCATIONS:
Overall Officials: Satu-Liisa K Pauniaho, MD, PhD, Principal Investigator — Tampere University Hospital, Finland
Locations (1):
- Tampere University Hospital, Tampere, Finland